CLINICAL TRIAL: NCT00312104
Title: Comparison of Efficacy and Safety of Insulin Detemir and Insulin Glargine in Patients With Type 1 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1372
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin glargine
Drug: insulin aspart

SUMMARY:
The trial is conducted in Europe and Africa. The aim of the trial is to compare the use of insulin detemir twice daily combined with mealtime insulin aspart against that of insulin glargine once daily combined with mealtime insulin aspart. The trial involves patients with Type 1 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Current daily insulin dose of more than 1.4 IU/kg
* BMI lesser than or equal to 35 kg/m2
* HbA1c greater than 7.5% and less than or equal to 12.0%
* In Austria, age more than 19 years

Exclusion Criteria:

* Proliferate retinopathy or maculopathy
* Recurrent major hypoglycaemia
* Any condition or disease such as uncontrolled hypertension or AIDS/HIV that rule out trial participation according to the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2002-04; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 26 weeks of treatment

SECONDARY OUTCOMES:
Adverse events
Body weight
Blood glucose
Hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (42):
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Vienna
- Germany (37):
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Diez
  - Novo Nordisk Investigational Site, Erlangen
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Flensburg
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Genthin
  - Novo Nordisk Investigational Site, Halle
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Heidelberg
  - Novo Nordisk Investigational Site, Hennigsdorf
  - Novo Nordisk Investigational Site, Hünxe
  - Novo Nordisk Investigational Site, Jena
  - Novo Nordisk Investigational Site, Kiel
  - Novo Nordisk Investigational Site, Landau
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Marl
  - Novo Nordisk Investigational Site, Mönchengladbach
  - Novo Nordisk Investigational Site, Neunkirchen
  - Novo Nordisk Investigational Site, Neuss
  - Novo Nordisk Investigational Site, Northeim
  - Novo Nordisk Investigational Site, Nuremberg
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Rheda-Wiedenbrück
  - Novo Nordisk Investigational Site, Saarbrücken
  - Novo Nordisk Investigational Site, Saarlouis
  - Novo Nordisk Investigational Site, Schönebeck
  - Novo Nordisk Investigational Site, Schwabenheim
  - Novo Nordisk Investigational Site, Schwerin
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wiesbaden
  - Novo Nordisk Investigational Site, Würzburg
- South Africa (3):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape

REFERENCES:
- [Result] Pieber TR, Treichel HC, Hompesch B, Philotheou A, Mordhorst L, Gall MA, Robertson LI. Comparison of insulin detemir and insulin glargine in subjects with Type 1 diabetes using intensive insulin therapy. Diabet Med. 2007 Jun;24(6):635-42. doi: 10.1111/j.1464-5491.2007.02113.x. Epub 2007 Mar 22. PMID 17381500
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com